CLINICAL TRIAL: NCT03573765
Title: The Role of Patient Factors, Surgical Factors and Hospital Factors Upon Patient Outcomes and NHS Costs in the Treatment of Upper Limb Musculoskeletal Conditions: Spatial and Iongitudinal Analysis of Routine Data
Brief Title: Epidemiology and Outcomes of Upper Limb Surgery: Analysis of Routine Data
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Arthritis Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: 12787; DARS-NIC-29827-Q8Z7Q (Other: NHS Digital)
Record Dates: First submitted 2018-06-04; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis; Dislocations; Inflammatory Arthritis; Rotator Cuff Tear; Shoulder Dislocation; Upper Limb Nerve Lesion; Shoulder Arthropathy; Elbow Arthropathy; Wrist Arthropathy; Arthropathy Unspecified, Involving Hand; Fracture, Shoulder; Fracture Elbow; Fracture Wrist and Hand; Dupuytren Contracture; Impingement Syndrome, Shoulder; Trigger Digit; Avascular Necrosis
Keywords: epidemiology; upper limb; hand surgery; wrist surgery; shoulder surgery; elbow surgery; outcomes; complications; revision surgery
MeSH Terms: conditions — Osteoarthritis; Joint Dislocations; Arthritis; Rotator Cuff Injuries; Shoulder Dislocation; Joint Diseases; Shoulder Fractures; Elbow Fractures; Wrist Fractures; Dupuytren Contracture; Shoulder Impingement Syndrome; Trigger Finger Disorder; Osteonecrosis | interventions — Arthroplasty, Replacement, Shoulder; Arthroplasty, Replacement, Elbow; Injections, Intra-Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Shoulder arthroplasty — Any form of joint replacement of the glenohumeral joint including prosthetic and excision.
Procedure: Elbow arthroplasty — Any form of joint replacement of the elbow joint including prosthetic and excision.
Procedure: Hand and wrist arthroplasty — Any form of joint replacement of joints of the hand and wrist including prosthetic and excision.
Procedure: Nerve decompression — Open or endoscopic release of peripheral nerve entrapment - subdivided by anatomical site of compression. Specific subgroups will include carpal tunnel and cubital tunnel release.
Procedure: Tendon repair — Open or arthroscopic repair or reconstruction of tendons of the shoulder, hand and upper limb in general.
Procedure: Joint stabilisation — Any procedure designed to increase stability of a joint, including soft tissue and bony blocking procedures.
Procedure: Excision/division/release of palmar fascia — Any procedure performed for treatment of Dupuytren's contracture.
Procedure: Surgical fixation of fractures — Any internal or external fixation of upper limb fractures - analysed by anatomical site.
Procedure: Soft tissue release/debridement/excision — Any removal or release of soft tissue for treatment of stiffness, functional impairment or pain. Specific subgroups will include trigger finger release, subacromial surgery and surgery for frozen shoulder.
Procedure: Intra-articular injection — Any intra-articular injection

SUMMARY:
Surgery is a common treatment type for damaged joints, tendons and nerves in the upper limb where conservative measures are inappropriate or have failed. These conditions are common and result in significant levels of pain and functional disability. The investigators are conducting a broad ranging study of variation in the provision of surgical treatment and factors affecting outcomes after surgical treatment of upper limb conditions. This will be a population-based study of all patients undergoing surgical treatment funded by the National Health Service (NHS) of England over a nineteen-year period. This study will help to understand the factors associated with a poor outcome following surgery, which can be shared with patients considering treatment options. The investigators will also document current and future health service burden associated with commonly performed surgical procedures including complications and repeat operations.

DETAILED DESCRIPTION:
The investigators will conduct time series analyses, geospatial mapping and risk-factor association studies for both access to and outcomes of surgical treatments of the upper limbs. A large cohort of pseudonymised records will be extracted from the NHS Hospital Episode Statistics Admitted Patient Care database. Suitable patients will be identified based on a match to a specified list of International Classification of Diseases (ICD-10) and Office for Population Censuses and Surveys (OPCS-4) codes. Dates and cause of death will be linked from the Office for National Statistics (ONS) by NHS Digital.

Separate analyses will be conducted for different intervention types with detailed outcomes reporting for high volume procedures. Adults will be defined as those aged 18 years or older at the time of surgery. Children will be defined as those aged less than 18 years at surgery and only included in a limited number of analyses where relevant (e.g. trigger digit).

Key analyses:

1. Baseline demographics by procedure type
2. Procedure volume incidence trends

   * Time series analysis
   * Adjusted to standard population distributions
   * Geographical mapping including adjustment for sociodemographic indices including indices of deprivation
3. Revision, reoperation and mortality rates:

   * Estimation by Kaplan Meier and actuarial life table methods
   * Life time risk calculated by the cumulative probability method
   * Cox regression adjusted for comorbidities and demographic, social and geographic factors
4. Complications, length of stay, costs:

   * Logistic and linear regression models for binary and continuous outcomes respectively
   * Adjusted for comorbidities and demographic, social and geographic factors

Where appropriate, the impact of replacing missing data will be explored with use of multiple imputation. All suitable patients will be entered into analyses to maximise statistical efficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Condition affecting one of:

   * Shoulder
   * Elbow
   * Wrist
   * Hand

   AND
2. All patients treated with surgery for any of the following:

   * Osteoarthritis
   * Inflammatory arthritis
   * Any other cause of arthropathy
   * Tendon tears
   * Peripheral neuropathy
   * Fractures and/or dislocations
   * Instability

   OR
3. Any arthroplasty surgery using a prosthesis

Exclusion Criteria:

* Patients registering a "type 2 opt out" - withholding NHS data from research use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing treatment funded by or in NHS hospitals in England and recorded in the Hospital Episode Statistics Admitted Patient Care database.
Sampling Method: Non-Probability Sample
Enrollment: 8308821 (Actual)
Dates: Start 1998-04-06 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Revision and reoperation | 1998-2017
  Estimated at annual increments and standardised lifetime risk
Treatment volume: time series | 1998-2017
  Crude and adjusted for population by age/sex
Treatment volume: geospatial patterns | 1998-2017
  Mapped according to residence and NHS organisation boundaries

SECONDARY OUTCOMES:
Complications | 30, 45, 60, 90 days post surgery + 1 year and last recorded follow-up/censoring.
  Death and infection for all. Specific adverse events dependent on procedure, e.g. periprosthetic fracture after arthroplasty surgery
Length of stay post surgery | up to 52 weeks from date of surgery
  Number of days - defined by time elapsed between surgery and the end of NHS spell.
Readmission to hospital | up to 30 days following surgery
  Number of patients readmitted to acute NHS trust
Healthcare related costs | up to 52 weeks from date of surgery
  Calculated from Healthcare Resource Group codes for index episode and related episodes

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Furniss, DPhil, Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rees JL, Craig R, Nagra N, Baldwin M, Lane JCE, Price A, Beard DJ, Abram S, Judge A, Prieto-Alhambra D, Furniss D, Carr AJ. Serious adverse event rates and reoperation after arthroscopic shoulder surgery: population based cohort study. BMJ. 2022 Jul 6;378:e069901. doi: 10.1136/bmj-2021-069901. PMID 35938625
- [Derived] Alser O, Abram SGF, Craig RS, Lane JCE, Shaw AV, Prats-Uribe A, Rees JL, Prieto-Alhambra D, Furniss D. Temporal Trends and Geographical Variation in Dupuytren Disease Surgery in England: A Population-Based Cohort Study. Ann Plast Surg. 2021 Sep 1;87(3):265-270. doi: 10.1097/SAP.0000000000002734. PMID 34397515
- [Derived] Lane JC, Craig R, Rees JL, Gardiner M, Mikhail MM, Riley N, Prieto-Alhambra D, Furniss D. Low rates of serious complications and further procedures following surgery for base of thumb osteoarthritis: analysis of a national cohort of 43 076 surgeries. BMJ Open. 2021 Jul 7;11(7):e045614. doi: 10.1136/bmjopen-2020-045614. PMID 34233971
- [Derived] Lane JCE, Craig RS, Rees JL, Gardiner MD, Shaw AV, Spiteri M, Kuo R, Dean BF, Green J, Prieto-Alhambra D, Furniss D. Low rate of subsequent surgery and serious complications following intra-articular steroid injection for base of thumb osteoarthritis: national cohort analysis. Rheumatology (Oxford). 2021 Sep 1;60(9):4262-4271. doi: 10.1093/rheumatology/keaa925. PMID 33410485
- [Derived] Lane JCE, Craig RS, Rees JL, Gardiner MD, Green J, Prieto-Alhambra D, Furniss D. Serious postoperative complications and reoperation after carpal tunnel decompression surgery in England: a nationwide cohort analysis. Lancet Rheumatol. 2020 Sep 30;3(1):e49-e57. doi: 10.1016/S2665-9913(20)30238-1. eCollection 2021 Jan. PMID 33381769
- [Derived] Craig RS, Lane JCE, Carr AJ, Furniss D, Collins GS, Rees JL. Serious adverse events and lifetime risk of reoperation after elective shoulder replacement: population based cohort study using hospital episode statistics for England. BMJ. 2019 Feb 20;364:l298. doi: 10.1136/bmj.l298. PMID 30786996